CLINICAL TRIAL: NCT00263133
Title: Modulation of Visually Evoked Potentials by an Antidepressant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEP-1; EudraCT 2005-005417-37
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-05

CONDITIONS: Depression
Keywords: Depression; SSRI; Sertraline; synaptic plasticity; visually evoked potentials
MeSH Terms: conditions — Depression | interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline

SUMMARY:
12 normal healthy controls will be treated with 50 mg sertraline once daily for three weeks. Early amplitudes of visually evoked potentials will be examined at day 0, 10 and 21 and statistically compared. This study aims to examine a putative modulation of synaptic transmission and plasticity by an antidepressant and is part of a series of studies in healthy individuals and depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals 18-65 years

Exclusion Criteria:

* history of affective oder other psyhiatric disorder
* severe medical condition
* pregnancy or ineffective contraception
* active illicit drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-12; Study Completion 2006-01

PRIMARY OUTCOMES:
Amplitudes and latencies of early visually evoked potentials.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Normann, MD, Principal Investigator — Dept. of Psychiatry, University of Freiburg
Locations (1):
- Dept. of Psychiatry, University of Freiburg, Freiburg im Breisgau, Germany